CLINICAL TRIAL: NCT02585986
Title: Randomized, Double Blind, Placebo-controlled Intervention Study to Evaluate Safety and Efficiency of a Probiotic in Symptoms Reduction and Use of Topic Corticoids in Mild Atopic Dermatitis Patients Aged 4 to 17 Years
Brief Title: Intervention Study to Evaluate a Probiotic in Mild Atopic Dermatitis Young Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biopolis S.L. (Industry)
Collaborators: Korott, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATO/PRO1
Record Dates: First submitted 2015-10-13; First posted 2015-10-26 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): daily intake of 1 capsule containing probiotic.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): daily intake of 1 capsule containing placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — daily intake of 1 capsule probiotic
  Other Names: Active formulation
  Arms: Probiotic
Dietary Supplement: Placebo — daily intake of 1 capsule containing placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the beneficial effect of a probiotic preparation with an antiinflammatory and modulating activity on immunological processes, with positive results on different inflammatory and atopic conditions.

DETAILED DESCRIPTION:
In this study the investigators evaluate the safety and efficacy of a probiotic formulation in the reduction of symptoms and use of topic and systemic corticosteroids and antihistamines in the treatment of mild atopic dermatitis according to Hanifin and Rajka diagnostic criteria for atopic dermatitis, with a SCORAD (Scoring Atopic Dermatitis) index of 20 to 40, in patients 4 to 18 years old, that require the use of said drugs due to disease flare-ups, and to whom the usage of topic corticoids to control said flare-ups is indicated.

ELIGIBILITY:
Inclusion Criteria:

* patients that are 4 to 17 years of age.
* Patients diagnosed of atopic dermatitis according to Hanifin and Rajka diagnostic criteria for atopic dermatitis.
* Patients with a SCORAD score ranging from 20 to 40.
* Patients that are actually using, or in which the use of topic corticosteroids to treat the atopic dermatitis flare-ups.
* Patients whose parents or legal representative have signed the informed consent. If the patient is 12 year old or older, the patient has to sign a consent to enter the trial.

Exclusion Criteria:

* Pregnancy.
* Breastfeeding.
* Women of childbearing age that do not make a commitment to use any effective contraceptive method.
* Phototherapy treatments to atopic dermatitis
* Systemic corticoid therapy in the last two months.
* Immunosuppressive or cytostatic treatment in the last two months.
* Probiotic treatment in the last two months.
* Systemic antibiotic in the last four months.
* Fever (axillary temperature > 37ºC or equivalent)
* Severe allergic diseases-
* Immunodeficiency or cancer related processes.
* Other dermatological pathologies that could difficult the atopic dermatitis evaluation, or that require the continued use of topic corticosteroids.
* Any contraindication to any product or drug used during the trial, according to their technical files.
* Participation in any drug clinical trial in the last 3 months.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Time of use of topic corticosteroids | twelve weeks
  Duration of treatment with topic corticosteroids
Variation in SCORAD score during treatment | twelve weeks

SECONDARY OUTCOMES:
Variation in the Global Clinical Impression (CGI) score during treatment | twelve weeks
Exposure to other treatments | twelve weeks
  Duration of treatment with systemic corticosteroids or antihistamine drugs
side effects due to treatment in two arms of treatment | twelve weeks
  Number of side effects due to probiotic and due to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Navarro-López, MD, Principal Investigator — Universidad Católica San Antonio de Murcia; Ana A. Ramirez-Boscá, MD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Centro Dermatologico Estetico de Alicante, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ellis C, Luger T, Abeck D, Allen R, Graham-Brown RA, De Prost Y, Eichenfield LF, Ferrandiz C, Giannetti A, Hanifin J, Koo JY, Leung D, Lynde C, Ring J, Ruiz-Maldonado R, Saurat JH; ICCAD II Faculty. International Consensus Conference on Atopic Dermatitis II (ICCAD II): clinical update and current treatment strategies. Br J Dermatol. 2003 May;148 Suppl 63:3-10. doi: 10.1046/j.1365-2133.148.s63.1.x. No abstract available. PMID 12694268
- [Background] Leung DY, Bieber T. Atopic dermatitis. Lancet. 2003 Jan 11;361(9352):151-60. doi: 10.1016/S0140-6736(03)12193-9. PMID 12531593
- [Background] Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94. doi: 10.1056/NEJMra074081. No abstract available. PMID 18385500
- [Background] Levy RM, Gelfand JM, Yan AC. The epidemiology of atopic dermatitis. Clin Dermatol. 2003 Mar-Apr;21(2):109-15. doi: 10.1016/s0738-081x(02)00360-7. No abstract available. PMID 12706328
- [Background] Su JC, Kemp AS, Varigos GA, Nolan TM. Atopic eczema: its impact on the family and financial cost. Arch Dis Child. 1997 Feb;76(2):159-62. doi: 10.1136/adc.76.2.159. PMID 9068310
- [Background] Simpson EL, Hanifin JM. Atopic dermatitis. J Am Acad Dermatol. 2005 Jul;53(1):115-28. doi: 10.1016/j.jaad.2005.01.130. No abstract available. PMID 15965431
- [Background] Boguniewicz M, Leung DY. 10. Atopic dermatitis. J Allergy Clin Immunol. 2006 Feb;117(2 Suppl Mini-Primer):S475-80. doi: 10.1016/j.jaci.2005.10.018. PMID 16455350
- [Background] Ridao M. Dermatitis atópica: clínica, diagnóstico diferencial y tratamiento. Pediatr Integral 2004:8:204-10.
- [Background] Hanifin JM, Rajka G. Diagnosis features of atopic dermatitis. Acta Derm Venereol 1980;92:44-7.
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Sprikkelman AB, Tupker RA, Burgerhof H, Schouten JP, Brand PL, Heymans HS, van Aalderen WM. Severity scoring of atopic dermatitis: a comparison of three scoring systems. Allergy. 1997 Sep;52(9):944-9. doi: 10.1111/j.1398-9995.1997.tb01255.x. PMID 9298180
- [Background] Charman C, Williams H. Outcome measures of disease severity in atopic eczema. Arch Dermatol. 2000 Jun;136(6):763-9. doi: 10.1001/archderm.136.6.763. PMID 10871941
- [Background] Pucci N, Novembre E, Cammarata MG, Bernardini R, Monaco MG, Calogero C, Vierucci A. Scoring atopic dermatitis in infants and young children: distinctive features of the SCORAD index. Allergy. 2005 Jan;60(1):113-6. doi: 10.1111/j.1398-9995.2004.00622.x. PMID 15575941
- [Background] Bhor U, Pande S. Scoring systems in dermatology. Indian J Dermatol Venereol Leprol. 2006 Jul-Aug;72(4):315-21. doi: 10.4103/0378-6323.26722. No abstract available. PMID 16880586
- [Background] National Institute for health and clinical excellence. Atopic eczema in children. Management of atopic eczema in children from birth up to the age of 12 years. NICE clinical guideline 57. Dec 2007.
- [Background] Boguniewicz M, Schmid-Grendelmeier P, Leung DY. Atopic dermatitis. J Allergy Clin Immunol. 2006 Jul;118(1):40-3. doi: 10.1016/j.jaci.2006.04.044. Epub 2006 Jun 6. No abstract available. PMID 16815136
- [Background] Schoepe S, Schacke H, May E, Asadullah K. Glucocorticoid therapy-induced skin atrophy. Exp Dermatol. 2006 Jun;15(6):406-20. doi: 10.1111/j.0906-6705.2006.00435.x. PMID 16689857
- [Background] Castro AP. Calcineurin inhibitors in the treatment of allergic dermatitis. J Pediatr (Rio J). 2006 Nov;82(5 Suppl):S166-72. doi: 10.2223/JPED.1557. PMID 17136292
- [Background] Meurer M, Folster-Holst R, Wozel G, Weidinger G, Junger M, Brautigam M; CASM-DE-01 study group. Pimecrolimus cream in the long-term management of atopic dermatitis in adults: a six-month study. Dermatology. 2002;205(3):271-7. doi: 10.1159/000065863. PMID 12399676
- [Background] Meurer M, Fartasch M, Albrecht G, Vogt T, Worm M, Ruzicka T, Altmeyer PJ, Schneider D, Weidinger G, Braeutigam M; CASM-DE-01 Study Group. Long-term efficacy and safety of pimecrolimus cream 1% in adults with moderate atopic dermatitis. Dermatology. 2004;208(4):365-72. doi: 10.1159/000078462. PMID 15178928
- [Background] de Benedictis FM, de Benedictis D, Canonica GW. New oral H1 antihistamines in children: facts and unmeet needs. Allergy. 2008 Oct;63(10):1395-404. doi: 10.1111/j.1398-9995.2008.01771.x. PMID 18782118
- [Derived] Climent E, Martinez-Blanch JF, Llobregat L, Ruzafa-Costas B, Carrion-Gutierrez MA, Ramirez-Bosca A, Prieto-Merino D, Genoves S, Codoner FM, Ramon D, Chenoll E, Navarro-Lopez V. Changes in Gut Microbiota Correlates with Response to Treatment with Probiotics in Patients with Atopic Dermatitis. A Post Hoc Analysis of a Clinical Trial. Microorganisms. 2021 Apr 15;9(4):854. doi: 10.3390/microorganisms9040854. PMID 33921166
- [Derived] Navarro-Lopez V, Ramirez-Bosca A, Ramon-Vidal D, Ruzafa-Costas B, Genoves-Martinez S, Chenoll-Cuadros E, Carrion-Gutierrez M, Horga de la Parte J, Prieto-Merino D, Codoner-Cortes FM. Effect of Oral Administration of a Mixture of Probiotic Strains on SCORAD Index and Use of Topical Steroids in Young Patients With Moderate Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jan 1;154(1):37-43. doi: 10.1001/jamadermatol.2017.3647. PMID 29117309